CLINICAL TRIAL: NCT03029052
Title: A Comparative Pilot Study in an Infectious Disease Department Assessing the Impact of Medication Reconciliation at Discharge Associated With a Patient's Counseling Session, Both Provided by a Pharmacist, on Patient's Care After Discharge
Brief Title: Medication Reconciliation at Discharge: Impact on Patient's Care
Acronym: CONCIVILLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Frederique Bouchand, PharmD, Centre d'Investigation Clinique et Technologique 805
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01628-43
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Medication Reconciliation
MeSH Terms: interventions — Medication Reconciliation

STUDY DESIGN:
Intervention Model Description: Monocenter, randomized, controlled, pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Medical and pharmaceutical management (at admission, during hospitalization and at discharge) will follow standard healthcare procedures of the department.
- Reconciliation group (Experimental): Standard healthcare procedures and pharmacist's involvement
  Interventions: Behavioral: Reconciliation

INTERVENTIONS:
Behavioral: Reconciliation — In addition to standard healthcare procedures, the pharmacist will analyze discharge prescriptions and proceed to medication reconciliation. A patient's counseling session will also be provided by the pharmacist. A reconciliation mail will be addressed to the PCP.
  Arms: Reconciliation group

SUMMARY:
Patient's discharge from hospital is associated with iatrogenic events for 12 to 17% of patients. This risk may be linked with discontinuity of care between hospital physicians and Primary Care Physician (PCP). The investigators aim to assess in this study the impact of medication reconciliation at discharge associated with a patient's counseling session, both provided by a pharmacist, on patient's care after discharge. To demonstrate the interest of medication reconciliation at discharge we expect a reduction by 15% of the number of prescription changes not maintained by the PCP after discharge.

DETAILED DESCRIPTION:
Patient's discharge from hospital is associated with iatrogenic events for 12 to 17% of patients and may lead to further hospitalization. This risk may be linked with discontinuity of care between hospital physicians and Primary Care Physician (PCP) and from discrepancies between patient's current medications and drugs prescribed at discharge.

Preventing adverse drug events (ADEs) remains a patient safety priority not only in hospitals but also across the continuum of care for patients. Implementing medication reconciliation at all transitions in care is an effective strategy for preventing discrepancies and ADEs. Medication reconciliation prevents and corrects medication errors by promoting transmissions of complete and accurate information about medicines.

Furthermore, ADEs may be the result of a failure to understand and manage post-discharge care needs and can lead to hospital readmission.

We assume that medication reconciliation at discharge, secondarily transmitted to the PCP with a discharge counseling session between the patient and a clinical pharmacist could have a positive impact on the maintenance of therapeutic optimization decided by in-hospital practitioners.

In order to evaluate this assumption, we will conduct a randomized controlled study on 120 patients (as a reduction by 15% of the number of prescription changes not maintained by the PCP after discharge is expected).

The follow-up will last 1 month after discharge from hospital. The first prescription from the PCP will be collected and analyzed. In addition, patients and PCPs will be contacted by the pharmacist to answer specific questionnaires.

The primary objective of the study is to assess the impact of medication reconciliation at discharge associated with a patient's counseling session, both provided by a pharmacist, on patient's care after discharge.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* hospitalized in infectious disease department
* with a chronic disease and a current medical prescription including at least three drugs
* discharged home or nursing home
* not opposed to the study

Exclusion Criteria:

* foreigners, patients under legal guardianship
* advanced dementia (MMS<20) or phone tracking impossible
* primary care physician opposed to answer questionnaire

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Proportion of in-hospital prescription changes not maintained by the Primary Care Physician (PCP) one month after discharge. | 1 month
  The number of in-hospital prescription changes will be evaluated only on discharge prescription transmitted to the patient (after prescription analysis by a clinical pharmacist in the "reconciliation" group)
  Compared to the list of all current medications at admission, in-hospital prescription changes include the following:
  * Adding a new drug
  * Discontinuing a drug
  * Drug switch
  * Modifying a dose
  Among these hospital prescription changes, some will not be maintained by the PCP one month after discharge.
  In-hospital prescription changes not maintained by the PCP will be evaluated on the first prescription of the PCP following discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Frederique BOUCHAND, PharmD, Principal Investigator — APHP; Benjamin DAVIDO, MD, Study Director — APHP
Locations (1):
- Hôpital Raymond poincaré, Garches, France

IPD SHARING:
Plan to Share IPD: No